CLINICAL TRIAL: NCT02994394
Title: A Study of OPC-41061 Orally Disintegrating (OD) Tablets Using 2 Different Formulations and 2 Dosing Regimens in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 156-102-00136; JapicCTI-163471 (Other: Japic)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Healthy Adult Male
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- OPC41061(15 mg) disintegrating tablet with water (Experimental): OPC41061 (15 mg) orally disintegrating tablet is administered with water.
  Interventions: Drug: OPC-41061
- OPC-41061(15 mg) disintegrating tablet without water (Experimental): OPC41061 (15 mg) orally disintegrating tablet is administered without water.
  Interventions: Drug: OPC-41061
- OPC-41061(15 mg) conventional tablet with water (Experimental): OPC-41061 (15 mg) conventional tablet is administered with water.
  Interventions: Drug: OPC-41061
- OPC41061(30 mg) disintegrating tablet with water (Experimental): OPC41061 (30 mg) orally disintegrating tablet is administered with water.
  Interventions: Drug: OPC-41061
- OPC-41061(30 mg) disintegrating tablet without water (Experimental): OPC41061 (30 mg) orally disintegrating tablet is administered without water.
  Interventions: Drug: OPC-41061
- OPC-41061(30 mg) conventional tablet with water (Experimental): OPC-41061 (30 mg) conventional tablet is administered with water.
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061

SUMMARY:
To assess the bioequivalence of OPC-41061 OD tablets and OPC-41061 conventional tablets at 15 and 30 mg in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of at least 50.0 kg
* BMI [body weight in kg / (height in m)2] of at least 17.6 kg/m2 and less than 25.0 kg/m2
* Judged by the investigator or subinvestigator to be capable of providing written informed consent prior to the start of any trial-related procedures and capable of complying with the trial procedures for this study.

Exclusion Criteria:

* Judged by the investigator,subinvestigator, or sponsor to have a clinically significant abnormality in results of the screening examination (including a notable deviation from the site's standard values) or a medical history that could place the subject at risk or affect the evaluation of drug absorption, distribution, metabolism, or excretion
* History of alcohol or drug dependence or abuse within 2 years prior to the trial
* History or current infection with hepatitis or acquired immunodeficiency syndrome (AIDS) or carrier of hepatitis B positive surface antigen (HBsAg), anti-hepatitis C virus (HCV), human immunodeficiency virus (HIV), or syphilis based on the results of the Treponema pallidum (TP) antibody test or rapid plasma reagin (RPR) test
* History of any severe drug allergy
* Positive results in alcohol screening test or urine drug screening test at time of screening examination or trial site admission
* Use of any other investigational medicinal product (IMP) within 120 days prior to Period 1 IMP administration
* Consumption of any food or beverage containing St. John's wort within 14 days prior to Period 1 IMP administration
* Consumption of any food or beverage containing grapefruit, Seville orange, or star fruit within 7 days prior to Period 1 IMP administration
* Judgment by the investigator or subinvestigator that the subject should not participate in the study for any other reason.

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kyusyu Region, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center, open-label, randomized, 3-period 3-way, crossover study using 2 different formulations and 2 different dosing regimens investigated bioequivalence between tolvaptan orally disintegrating (OD) and conventional tablets in 84 healthy adult male subjects in 2 cohorts. Bioequivalence between the OD and conventional 15 mg tablets was investigated in Cohort 1. In Cohort 2, bioequivalence between the OD and conventional 30 mg tablets was investigated.
Pre-assignment Details: A total of 84 subjects were divided into 2 cohorts of 42 subjects each. The 42 subjects each in 2 cohorts were randomly assigned to the conventional tablet first group, OD tablet with water first group, or OD tablet without water first group according to the randomization code in a 1:1:1 ratio. Forty subjects in Cohort 1 and 41 subjects in Cohort 2 completed the trial.
Groups:
- Cohort 1: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water; Cohort 1: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water; Cohort 1: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet: Subjects received single oral administration of tolvaptan 15 mg in Cohort 1, conventional or OD tablet, with or without water on each administration day in Period 1, Period 2, and Period 3.
  A washout period of 72 hours was set from postdose in Period 1 until predose in Period 2 and from postdose in Period 2 until predose in Period 3.
- Cohort 2: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water; Cohort 2: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water; Cohort 2: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet: Subjects received single oral administration of tolvaptan 30 mg in Cohort 2, conventional or OD tablet, with or without water on each administration day in Period 1, Period 2, and Period 3.
  A washout period of 72 hours was set from postdose in Period 1 until predose in Period 2 and from postdose in Period 2 until predose in Period 3.
Period: Period 1 (Days 1 to 3)
Arm/Group | Cohort 1: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water | Cohort 1: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water | Cohort 1: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet | Cohort 2: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water | Cohort 2: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water | Cohort 2: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet
Started | 14 | 14 | 14 | 14 | 14 | 14
Completed | 14 | 14 | 13 | 14 | 14 | 14
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2 (Days 4 to 6)
Arm/Group | Cohort 1: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water | Cohort 1: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water | Cohort 1: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet | Cohort 2: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water | Cohort 2: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water | Cohort 2: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet
Started | 14 | 14 | 13 | 14 | 14 | 14
Completed | 14 | 13 | 13 | 14 | 13 | 14
Not Completed | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0
Period: Period 3 (Days 7 and 8)
Arm/Group | Cohort 1: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water | Cohort 1: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water | Cohort 1: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet | Cohort 2: Conventional Tablet, Then OD Tablet Without Water, Then OD Tablet With Water | Cohort 2: OD Tablet With Water, Then Conventional Tablet, Then OD Tablet Without Water | Cohort 2: OD Tablet Without Water, Then OD Tablet With Water, Then Conventional Tablet
Started | 14 | 13 | 13 | 14 | 13 | 14
Completed | 14 | 13 | 13 | 14 | 13 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all subjects that received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Cohort 1: Subjects received single oral administration of tolvaptan 15 mg in Cohort 1, conventional or OD tablet, with or without water on each administration day in Period 1, Period 2, and Period 3.
  A washout period of 72 hours was set from postdose in Period 1 until predose in Period 2 and from postdose in Period 2 until predose in Period 3.
- Cohort 2: Subjects received single oral administration of tolvaptan 30 mg in Cohort 2, conventional or OD tablet, with or without water on each administration day in Period 1, Period 2, and Period 3.
  A washout period of 72 hours was set from postdose in Period 1 until predose in Period 2 and from postdose in Period 2 until predose in Period 3.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (4.3) | 23.5 (4.8) | 24.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 42 | 42 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 42 | 42 | 84
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Tolvaptan
Description: Blood sampling for plasma tolvaptan concentration before IMP administration and 1, 2, 3, 4, 5, 6, 8, 10, 12, and 16 hours postdose in each period in Cohort 1 and 2 was performed for pharmacokinetic evaluation.
Time Frame: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 hours post-dose
Population: Bioequivalence analysis set: all subjects with both AUCt and Cmax values across Period 1, Period 2, and Period 3.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1: 15 mg Conventional Tablet: Single oral administration of 1 tolvaptan 15 mg conventional tablet with water under fasting conditions
- Cohort 1: 15 mg OD Tablet Without Water: Single oral administration of 1 tolvaptan 15 mg OD tablet without water under fasting conditions
- Cohort 1: 15 mg OD Tablet With Water: Single oral administration of 1 tolvaptan 15 mg OD tablet with water under fasting conditions
- Cohort 2: 30 mg Conventional Tablet: Single oral administration of 1 tolvaptan 30 mg conventional tablet with water under fasting conditions
- Cohort 2: 30 mg OD Tablet Without Water: Single oral administration of 1 tolvaptan 30 mg OD tablet without water under fasting conditions
- Cohort 2: 30 mg OD Tablet With Water: Single oral administration of 1 tolvaptan 30 mg OD tablet with water under fasting conditions
Arm/Group | Cohort 1: 15 mg Conventional Tablet | Cohort 1: 15 mg OD Tablet Without Water | Cohort 1: 15 mg OD Tablet With Water | Cohort 2: 30 mg Conventional Tablet | Cohort 2: 30 mg OD Tablet Without Water | Cohort 2: 30 mg OD Tablet With Water
Number analyzed (Participants) | 39 | 39 | 39 | 41 | 41 | 41
ng/mL | 131 (71.0) | 149 (72.6) | 125 (63.1) | 203 (72.7) | 218 (56.0) | 198 (54.7)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Observable Concentration at Time t (AUCt) of of Tolvaptan
Description: as for outcome 1
Time Frame: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 hours post-dose
Population: Bioequivalence analysis set: all subjects with both AUCt and Cmax values across Period 1, Period 2, and Period 3.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: 15 mg Conventional Tablet | Cohort 1: 15 mg OD Tablet Without Water | Cohort 1: 15 mg OD Tablet With Water | Cohort 2: 30 mg Conventional Tablet | Cohort 2: 30 mg OD Tablet Without Water | Cohort 2: 30 mg OD Tablet With Water
Number analyzed (Participants) | 39 | 39 | 39 | 41 | 41 | 41
ng*h/mL | 697 (440) | 674 (361) | 685 (392) | 1120 (334) | 1130 (306) | 1110 (312)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected during the treatment period (8 days)
Description: Safety analysis set: all subjects that received at least 1 dose of IMP.
Arm/Group | Cohort 1: 15 mg Conventional Tablet | Cohort 1: 15 mg OD Tablet Without Water | Cohort 1: 15 mg OD Tablet With Water | Cohort 2: 30 mg Conventional Tablet | Cohort 2: 30 mg OD Tablet Without Water | Cohort 2: 30 mg OD Tablet With Water
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/41 | 0/42 | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/41 | 0/42 | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 1/41 | 1/41 | 2/41 | 1/42 | 0/42 | 0/41
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 15 mg Conventional Tablet (N=41) | Cohort 1: 15 mg OD Tablet Without Water (N=41) | Cohort 1: 15 mg OD Tablet With Water (N=41) | Cohort 2: 30 mg Conventional Tablet (N=42) | Cohort 2: 30 mg OD Tablet Without Water (N=42) | Cohort 2: 30 mg OD Tablet With Water (N=41)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT02994394/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT02994394/SAP_001.pdf